CLINICAL TRIAL: NCT00608543
Title: Aripiprazole Augmentation of SSRI Antidepressant Therapy in Treatment Refractory Depression: Assessment of Symptom Reduction, Psychosocial Function, and Cognitive Function
Brief Title: Aripiprazole Augmentation of SSRI Therapy in Treatment Refractory Depression
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Texas Southwestern Medical Center (Other)
Collaborators: Bristol-Myers Squibb (Industry)
Responsible Party: Principal Investigator, Prabha Sunderajan, Assistant Professor, University of Texas Southwestern Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 042004-011
Record Dates: First submitted 2008-01-23; First posted 2008-02-06 (Estimated); Results first posted 2012-10-26 (Estimated); Last update posted 2012-10-26 (Estimated); Status verified 2012-03

CONDITIONS: Major Depressive Disorder
Keywords: cognitive function; psychosocial function; augmentation; treatment refractory depression
MeSH Terms: conditions — Depressive Disorder, Major; Depressive Disorder, Treatment-Resistant | interventions — Aripiprazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Aripiprazole augmentation (Other): This is a single arm trial in which all participants recieved open label aripiprazole augmentation of their current escitalopram, citalopram or sertraline treatment.
  Interventions: Drug: Aripiprazole

INTERVENTIONS:
Drug: Aripiprazole — varied dose (5, 10, 15 mg qd) for 6 wks
  Other Names: Abilify

SUMMARY:
Our target population will have been adequately treated with one of three selective serotonin reuptake inhibitors (SSRIs; escitalopram, citalopram, or sertraline) for at least 8-12 weeks and continue to experience symptoms of depression that have prompted them to seek additional treatment. Escitalopram, citalopram, and sertraline were selected for use in this study because they are among the most commonly selected SSRIs and they are associated with a reduced likelihood of drug-drug interactions with aripiprazole. After completion of the screening process, eligible participants will be augmented with aripiprazole (5, 10, or 15 mg) for 6 weeks. Participants will continue SSRI treatment with their prescribing physician, in conjunction with study participation. Symptom severity will be assessed on a weekly basis, and cognitive and psychosocial function will be assessed at pre- and post-augmentation. We hypothesize that aripiprazole augmentation will be associated with reductions in symptom severity, and with improved performance on measures of psychosocial and cognitive function.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-65
* Primary diagnosis of Major Depressive Disorder (MDD)
* Completion of at least 8-12 weeks (and no longer than 6 months) of treatment with escitalopram, citalopram, or sertraline, with at least 6 weeks at an adequate dose (i.e., 20 mg escitalopram; 40 mg citalopram; 150 mg sertraline)
* Hamilton Rating Scale for Depression, 17-item (HRSD17) score less than or equal to 14 and/or Clinical Global Impression - Severity (CGI-S) score less than or equal to 3
* Self-reported difficulties with cognition and/or concentration, and an Inventory for Depressive Symptomatology Clinician-Rated, 30-item (IDS-C30) item #16 (Concentration and Decision Making) score less than or equal to 2
* Ability to read and write in English (required because instructions for cognitive testing and several questionnaires are available only in English)

Exclusion Criteria:

* Presence of untreated or unstable comorbid medical condition based on physician information or evidence at examination, such as hypertension, diabetes, hypothyroidism.
* Presence of known cardiovascular disease or seizure disorder.
* Presence of other primary psychiatric disorders or conditions (including depression due to medical conditions, currently suicidal or high suicide risk, current or past psychotic disorders of any type, bipolar disorder (I, II, or Not Otherwise Specified [NOS]), schizophrenia, schizoaffective disorder, anorexia, bulimia, obsessive compulsive disorder, alcohol or substance abuse or dependence within the last 6 months)
* Presence of organic brain injury or dementia, based on a cutoff score of < 20 on the Mini Mental Status Examination (MMSE).
* Concomitant pharmacological or psychotherapeutic treatment (in addition to one SSRI as described in Inclusion Criteria) including but not limited to anxiolytics, neuroleptics, mood stabilizers
* Hospitalization for mental illness within the past year.
* For women, currently pregnant or planning to become pregnant in the next year.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2005-10; Primary Completion 2009-01 (Actual); Study Completion 2009-01 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- University of Texas Southwestern Medical Center at Dallas, Dallas, Texas, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Open-label Aripiprazole Augmentation: Aripiprazole augmentation of existing escitalopram, citalopram, or sertraline treatment was provided to study participants at a flexible dose between 5-15 mg (based on clinical symptoms and side effects) for 6 weeks
Period: Overall Study
Arm/Group | Open-label Aripiprazole Augmentation
Started | 17
Completed | 13
Not Completed | 4
Not completed — Adverse Event | 4

BASELINE CHARACTERISTICS:
Arm/Group | Open-label Aripiprazole Augmentation
Number analyzed (Participants) | 17
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 17
  >=65 years | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 48.18 (7.95)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13
  Male | 4
Region of Enrollment [Number; unit: participants]
  United States | 17

OUTCOME MEASURES:

1. Primary Outcome: Stockings of Cambridge (SOC) Mean Initial Thinking Time for 3-move Problems
Description: The SOC is part of the CAmbridge Neuropsychological Test Automated Battery (CANTAB) and is an executive function task based on the Tower of London test that assesses spatial planning for problems with 2, 3, 4, or 5 moves. The Mean Initial Thinking Time for 3-move problems is the time (in milliseconds)taken to plan a problem solution for trials requiring 3 moves. Higher numbers indicate poorer performance. Time reported is the difference between baseline and 6 weeks post-treatment.
Time Frame: baseline and 6 weeks
Population: Completers; due to fact that testing occurred at pre- and post-intervention; mean represents difference between pre- and post-intervention
Measure: Mean (Standard Deviation); unit: milliseconds
Groups:
- Open Label Aripiprazole Augmentation: This is a single arm trial in which all participants recieved open label aripiprazole augmentation of their current escitalopram, citalopram or sertraline treatment.
Arm/Group | Open Label Aripiprazole Augmentation
Number analyzed (Participants) | 13
milliseconds | -4485.50 (6279.40)

2. Secondary Outcome: Quality of Life Enjoyment and Satisfaction Questionnaire
Description: The Q-LES-Q general activities is designed to measure subjective satisfaction and enjoyment, as opposed to function, in various domains including physical health, feelings, work, household duties, school/course work, leisure time activities, social relations, and general activities. The raw score is converted into a percent of the maximum possible score and range from 0 to 100. Higher scores indicate greater enjoyment and satisfaction.
Time Frame: 6 weeks
Population: Study completers who completed the Q-LES-Q pre- and post-intervention; mean represents mean difference from pre- to post-intervention
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Open Label Aripiprazole Augmentation
Number analyzed (Participants) | 12
units on a scale | 0.81 (0.48)

3. Secondary Outcome: Change in Hamilton Rating Scale for Depression (HRSD - 17-item)
Description: The HRSD 17-item scale is a clinician-administered rating scale designed to assess the severity of symptoms in patients diagnosed with depression. Scores range from 0 to 52, with higher scores indicating higher levels of depression severity.
Time Frame: 6 weeks
Population: Study completers who completed the HRSD pre- and post-intervention; mean represents mean difference from pre- to post-intervention
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Open Label Aripiprazole Augmentation
Number analyzed (Participants) | 12
units on a scale | -11.42 (4.50)

4. Primary Outcome: Stockings of Cambridge (SOC) Mean Initial Thinking Time for 5-move Problems
Description: The SOC is part of the CAmbridge Neuropsychological Test Automated Battery (CANTAB) and is an executive function task based on the Tower of London test that assesses spatial planning for problems with 2, 3, 4, or 5 moves. The Mean Initial Thinking Time for 5-move problems is the time (in milliseconds) taken to plan a problem solution for trials requiring 5 moves. Higher numbers indicate poorer performance. Time reported is the difference between baseline and 6 weeks post-treatment.
Time Frame: baseline and 6 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: milliseconds
Arm/Group | Open Label Aripiprazole Augmentation
Number analyzed (Participants) | 13
milliseconds | -4676.10 (8604.16)

5. Primary Outcome: Spatial Working Memory (SWM) Between Errors for 6-move Problems
Description: The SWM task is part of the CANTAB neruopsychological test battery and is an executive function task assessing retention and manipulation of items in working memory, with the ability for assessment of perseverative (redundant) errors. Between errors are times the subject revisits a box in which a token was previously found; errors are calculated for 4-, 6-, and 8-box trials. Higher numbers indicate poorer performance. Errors reported are the difference between baseline and 6 weeks post-treatment.
Time Frame: baseline and 6 weeks
Population: Completers because data were collected pre- and post-treatment
Measure: Mean (Standard Deviation); unit: number of errors
Groups:
- Spatial Working Memory Between Errors for 6-move Problems: This is a single arm trial in which all participants recieved open label aripiprazole augmentation of their current escitalopram, citalopram or sertraline treatment.
Arm/Group | Spatial Working Memory Between Errors for 6-move Problems
Number analyzed (Participants) | 13
number of errors | -4.00 (4.67)

6. Primary Outcome: Spatial Working Memory (SWM) Strategy Score
Description: The SWM task is part of the CANTAB neruopsychological test battery and is an executive function task assessing retention and manipulation of items in working memory, with the ability for assessment of perseverative (redundant) errors. The Strategy score represents the number of times a participant begins a search with the same box for 6- and 8-box problems. Minimum score is 8 and maximum score is 56. Higher numbers indicate poorer performance. Score reported is the difference between baseline and 6 weeks post-treatment.
Time Frame: baseline and 6 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Open Label Aripiprazole Augmentation
Number analyzed (Participants) | 13
units on a scale | -3.15 (4.52)

ADVERSE EVENTS:
Arm/Group | Open-label Aripiprazole Augmentation
Serious Adverse Events (participants affected / at risk) | 0/17
Other Adverse Events (participants affected / at risk) | 14/17
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Open-label Aripiprazole Augmentation (N=17)
diarrhea (Gastrointestinal disorders) | 8
constipation (Gastrointestinal disorders) | 8
dry mouth (Gastrointestinal disorders) | 6
nausea/vomiting (Gastrointestinal disorders) | 3
palpitations (Cardiac disorders) | 2
dizziness on standing (Cardiac disorders) | 3
chest pain (Cardiac disorders) | 2
rash (Skin and subcutaneous tissue disorders) | 2
increased perspiration (Skin and subcutaneous tissue disorders) | 6
itching (Skin and subcutaneous tissue disorders) | 1
dry skin (Skin and subcutaneous tissue disorders) | 1
headache (Nervous system disorders) | 14
tremors (Nervous system disorders) | 4
poor coordination (Nervous system disorders) | 6
dizziness (Nervous system disorders) | 5
blurred vision (Eye disorders) | 5
ringing in the ears (Ear and labyrinth disorders) | 6
difficulty urinating (Renal and urinary disorders) | 1
general malaise (General disorders) | 8
restlessness (Nervous system disorders) | 12
fatigue (General disorders) | 13
decreased energy (General disorders) | 10
painful urination (Renal and urinary disorders) | 1
frequent urination (Renal and urinary disorders) | 6
menstrual irregularity (Reproductive system and breast disorders) | 2
difficulty sleeping (Nervous system disorders) | 13
sleeping too much (Nervous system disorders) | 9
loss of sexual desire (Reproductive system and breast disorders) | 11
trouble achieving orgasm (Reproductive system and breast disorders) | 4
trouble with erections (Reproductive system and breast disorders) | 1
anxiety (Nervous system disorders) | 10
poor concentration (Nervous system disorders) | 3

LIMITATIONS AND CAVEATS:
Note that because this is an augmentation trial, reported AEs are due to combined treatment with escitalopram, citalopram, or sertraline AND aripiprazole.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No